CLINICAL TRIAL: NCT04786808
Title: Risk Factors for COVID-19 Mortality: a Prospective Observational Study
Brief Title: Risk Factors for COVID-19 Mortality
Acronym: RF-COVID
Status: Terminated | Type: Observational
Why Stopped: Not enough participants recruited (about 30% at october 2021).
Sponsor: Teodoro Marcianò (Other)
Responsible Party: Sponsor-Investigator, Teodoro Marcianò, Doctor of Medicine, Emergency Medicine Specialist, Azienda Unita Sanitaria Locale di Piacenza
Organization: Azienda Unita Sanitaria Locale di Piacenza (Other)
Other Study IDs: RF-COVID-AUSLPC
Record Dates: First submitted 2021-03-05; First posted 2021-03-08 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: COVID-19 Virus Infection; Population at Risk; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 pandemic has deeply burdened hospitals all over the world. A two-stage disease has been hypothesized due to quick worsening of clinical status after 7-10 days from the beginning of first symptoms, generally flu-like symptoms. Predicting clinical worsening could help to address major efforts towards higher risk patients.

During the last year most observational studies, generally retrospective, has been conducted, identifying some risk factors such as age, obesity, male gender, cardiovascular disease, COPD, diabetes etc.

The study goal is to collect systematically a variegate amount of clinical, biometric, laboratory and radiological data from patients admitted to the Emergency Medicine Ward of Piacenza Hospital (Italy), in order to prospectively analyze what characteristics are associated to higher risk of mortality.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the Emergency Medicine Ward from the Emergency Department of Piacenza Hospital (Italy)
* Confirmed COVID-19 diagnosis through molecular test obtained from nasal-pharyngeal swabs in the Emergency Department
* Age above 18

Exclusion Criteria:

* inability to obtain an informed consent due to neurological conditions.
* patient's refusal to sign the informed consent
* inability of researchers to recruit the patient in the first 24 hours from the admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ward from the Emergency Department are proposed to participate to the study.
  Patients admitted to the Emergency Medicine Ward have a COVID-19 pneumonia with respiratory failure at any stage of severity, with a PaO2/FiO2 ratio approximately between 100 and 300. Prevalence of severe cases changes according to the number of cases diagnosed in the community and consequently to the global number of admissions to the hospital. The study is intended to be conducted over a period of 1 year.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-11-07 (Actual); Study Completion 2021-11-07 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 28 days after admission
  Number of patients who die for any cause in the first 28 days after admission

SECONDARY OUTCOMES:
Need of invasive ventilation | 15 days after admission
  Number of patients who need invasive ventilation in the first 15 days after admission

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL di Piacenza, Piacenza, Emilia-Romagna, Italy